CLINICAL TRIAL: NCT04155294
Title: Re-Evaluation of Annual Cytology Using HPV Testing to Upgrade Prevention (REACH-UP): a Feasibility Study in Women Living With HIV
Brief Title: Re-Evaluation of Annual Cytology Using HPV Testing to Upgrade Prevention in Women Living With HIV
Acronym: REACH-UP
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: British HIV Association (BHIVA) (Unknown)
Responsible Party: Sponsor
Other Study IDs: IRAS Reference 259611
Record Dates: First submitted 2019-10-18; First posted 2019-11-07 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Cervical Cancer; HPV Infection; HIV Infections
Keywords: HPV infection; Women; HIV Infection; Cervical cancer; Screening
MeSH Terms: conditions — Uterine Cervical Neoplasms; Papillomavirus Infections; HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Mucosal cells obtained by a vaginal swabs will be stored in Microbiology lab before analysis. Specimens will be destroyed after the study analysis if performed according to local regulation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Current British HIV Association (BHIVA) guidelines recommend annual cervical screening (with a cervical smear) for women living with HIV (WLWH). NHS guidelines for women in England will, however, change soon. Women will initially be tested for human papilloma virus (HPV), a virus which causes virtually all cervical cancer. Only those who are infected with HPV will then undergo the smear testing. The BHIVA guidelines, however, taking the view that HIV infection (and its ability to weaken the immune system) increases the risk of persistent HPV infection and of cancer in those who are infected, consider safer for all WLWH to go straight to annual smear testing. Most WLWH in the UK are now receiving treatment which protects their immune system - this suggests that less WLWH could be HPV infected. The identification of a group of WLWH who could benefit from less frequent screening could improve quality of life, and allow the NHS to reduce unnecessary tests and costs. A large study is needed to collect robust evidence that would support changes to standard practice. Before investing huge resources, the investigators need to know if a study would be feasible, conducting a pilot study on 70 WLWH aged 25-64, regularly attending clinics for HIV care. Participants will be asked to complete an entry survey and they will undergo routine cervical smears (baseline and after 1 year). At baseline, after six months, and one year women will take their own vaginal swabs for the detection of HR-HPV. An exit questionnaire will be undertaken at the last visit.

DETAILED DESCRIPTION:
This pilot study will enrol 70 WLWH aged 25-64, with no history of cervical abnormalities attending 4 HIV clinics in the UK. Participants will be asked to complete an entry survey in which behavioural information, gynaecological and sexual history, will be collected, with the aim of characterising the study population for the risk factors of HPV infection. Women's attitude towards the current cervical screening and their view on a change to HPV testing will also be assessed. Participants' relevant clinical data will be collected form their medical notes. Women will be instructed to perform a self-taken vaginal swab for the detection of HR HPV while in clinic, and they will be reminded of the annual cervical smear (which can be offered in clinic or performed at their GP practice as per local policy). After six months, women will be asked to take another vaginal swab; this can be offered in clinic, during the regular HIV follow up, or can be sent via the post. Another sample for HR-HPV testing will be collected one year later, at the next routine HIV appointment. The annual smear test will be due and this will be offered in clinic or done at the GP practice, according to local policies. After this visit, an exit questionnaire will be undertaken to evaluate the acceptability of the study procedures.

ELIGIBILITY:
INCLUSION CRITERIA

* Women aged 25-64
* HIV diagnosis ≥ 6 months
* No previous diagnosis of CIN 2/3 and/or treatment for cervical dysplasia
* Last smear test done ≥1 year before baseline
* Able to speak and understand English
* Willing and able to provide informed consent

EXCLUSION CRITERIA

* Suspected or known invasive cervical malignancy
* Currently pregnant or breast-feeding
* Any other condition, which, in the opinion of the Investigator, would make participation in the study unsafe or interfere with interpretation of the study outcomes.

Ages: 25 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — gender at birth
Study Population: Women aged 25-64 years living with HIV for at least 6 months with annual cervical smear due, in accordance with national guidelines. The majority of HIV women >25 years in 2019 will not have been vaccinated against HPV.
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of HR HPV in WLWH aged 25-64 years in the UK | baseline
  HPV DNA detected by PCR on vaginal self-taken swab

SECONDARY OUTCOMES:
Rates of enrolment | baseline
  Proportion of eligible women on all the women attending the Clinic
Response rate to questionnaires | 1 year
  Proportion of questionnaires completed
Feasibility of self-sampling | 1 year
  Proportion of HR-HPV self-sample tests returned
Participants retention rate | 1 year
  Proportion of patients who complete the study procedures
Acceptability of study procedures including self-taken vaginal swabs | 1 year
  questionnaire containing closed and opened questions and visual scale from 0 to 100, higher score indicate a better outcome
Awareness of cervical cancer risk | baseline
  questionnaire containing closed and opened questions and visual scale from 0 to 100, where higher scores indicate a better outcome
Compliance to standard screening procedures | baseline
  questionnaire containing closed and opened questions and visual scale from 0 to 100, where higher scores indicate a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Paola Cicconi, Principal Investigator — University of Oxford
Locations (6):
- United Kingdom (6):
  - Oxford University Hospital NHS Foundation Trust, Oxford, Oxfordshire
  - Buckinghamshire Healthcare NHS Trust, High Wycombe
  - Royal Free Hospital Nhs Foundation Trust, London
  - GUY's AND ST THOMAS' NHS FOUNDATION TRUSTS, London
  - Milton Keynes University NHS Foundation Trust, Milton Keynes
  - ROYAL BERKSHIRE NHS FOUNDATION TRUST, Upton Hospital, Albert Street, Slough

IPD SHARING:
Plan to Share IPD: No